CLINICAL TRIAL: NCT01665885
Title: HAIS-SE (Hypothermia in Acute Ischemic Stroke - Surface Versus Endovascular Cooling): A Randomized Trial Comparing Surface Versus Endovascular Cooling in Awake Stroke Patients Treated With Thrombolysis
Brief Title: Hypothermia in Acute Ischemic Stroke - Surface Versus Endovascular Cooling (HAIS-SE)
Acronym: HAIS-SE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Heidelberg (Other)
Collaborators: ZOLL Circulation, Inc., USA (Industry)
Responsible Party: Principal Investigator, Dr. Sven Poli, MD MSc FESO, Dr. Sven Poli, Consultant Neurologist, Principal Investigator, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAIS-SE
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2013-06

CONDITIONS: Ischemic Stroke; Thrombolysis; Hypothermia
Keywords: hypothermia; induction of hypothermia; non invasive cooling; external cooling; surface cooling; endovascular cooling; cooling catheter; stroke; shivering; neuro monitoring; coagulation
MeSH Terms: conditions — Ischemic Stroke; Hypothermia; Stroke; Thrombosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Endovascular cooling (Active Comparator): Endovascular cooling using the cooling device ZOLL Thermogard XP with ZOLL Quattro cooling catheter
  Interventions: Device: ZOLL Thermogard XP
- Surface cooling (Active Comparator): Surface cooling using the cooling device BARD/Medivance Arctic Sun 5000 with BARD/Medivance Arctic Gel Pads
  Interventions: Device: BARD/Medivance Arctic Sun 5000
- Control group (No Intervention): Best medical treatment following international stroke guidelines

INTERVENTIONS:
Device: ZOLL Thermogard XP — Induction of hypothermia with 1L cold crystalloid infusions (0,9%NaCl or Ringer's solution). Cooling catheter placement at the earliest 30min after end of thrombolysis.
  Other Names: ZOLL Thermogard XP cooling device, ZOLL Circulation, Inc., USA; ZOLL Quattro cooling catheter, ZOLL Circulation, Inc., USA
  Arms: Endovascular cooling
Device: BARD/Medivance Arctic Sun 5000 — Induction of hypothermia with 1L cold crystalloid infusions (0,9%NaCl or Ringer's solution) and simultaneous start of surface cooling.
  Other Names: BARD/Medivance Arctic Sun 5000, C. R. Bard, Inc., USA; BARD/Medivance Arctic Gel Pads, C. R. Bard, Inc., USA
  Arms: Surface cooling

SUMMARY:
HAIS-SE is evaluating for the first time ever in a randomized controlled trial efficacy, tolerability, practicability and safety of endovascular versus surface cooling in awake stroke patients.

DETAILED DESCRIPTION:
Mild hypothermia improves outcome in patients with global cerebral ischemia after cardiac arrest. Via animal models hypothermia has been identified as the most promising neuroprotective therapy in focal cerebral ischemia as well. But the prove of clinical benefit in patients with acute ischemic stroke is still missing: Most likely due to the prolonged time window until hypothermia-induction (14 h) in previous studies. In addition, feasibility of the method through which hypothermia is applied is crucial for a broad implementation of hypothermia in stroke therapy. Surface versus endovascular cooling have never been compared in a prospective trial in awake stroke patients.

HAIS-SE is evaluating for the first time ever in a randomized controlled trial efficacy, tolerability, practicability and safety of endovascular versus surface cooling in awake stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke
* Intravenous thrombolysis within 4.5h from symptom onset
* Informed consent of the patient
* NIHSS score ≥ 2 and ≤ 20
* Age ≥ 18 and ≤ 90 years
* Placement of cooling catheter / cooling pads within 6h from symptom onset

Exclusion Criteria:

* (Expected) intubation (e.g. for interventional treatment)
* Pregnancy
* Body weight > 120kg
* Body height < 150cm
* Life-expectancy < 3 months
* Fever > 38.5°C at screening
* Known hematologic disease with increased risk of thrombosis (e.g. cryoglobulinemia, cold agglutinins, sickle cell anemia)
* Known vasospastic vascular disorder (e.g. Raynaud's phenomenon or thromboangiitis obliterans)
* Possible compression of the inferior vena cava (e.g. due to tumor) or vena cava filter
* Acute pulmonary embolism
* Acute myocardial infarction
* Severe cardiac insufficiency (NYHA ≥ III)
* Threatening ventricular dysrhythmia
* QTc-interval > 450ms
* Bradycardia < 50/min
* Sick-Sinus-Syndrom
* AV-block > I°
* Severe infection with bacteremia or sepsis ≤ 72h
* Severe renal (GFR < 30ml/min) or liver insufficiency (Child-Pugh C)
* Myopathy
* Known intolerance or allergy against acetaminophen, buspirone, clonidine, magnesium sulphate or pethidine.
* Treatment with MAO-inhibitors ≤ 14 days
* Acute closed-angle glaucoma

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Body core temperature | 0 to 48h
  Primary endpoint: Time to primary target body core temperature (34°C) after hypothermia-induction.

SECONDARY OUTCOMES:
Efficacy | 0 to 48h
  Secondary efficacy outcome measures include the amount of patients reaching the primary target body core temperature (34°C), the time-frame until reaching 35°C body core temperature, temperature stability during maintenance and rewarming.
Tolerability | 0 to 48h
  Tolerability outcome measures include a specific Hypothermia Participant Experience Questionnaire (HPEQ) and the Bedside Shivering Assessment Scale (BSAS) plus correlation with skin temperature, EMG and sNIRS.
Practicability | 0 to 48h
  Practicability outcome measures include a specific Hypothermia Nursing Staff Experience Questionnaire (HNEQ).
Safety | 0 to d90
  Safety outcome measures include the analysis of (severe) adverse events (e.g. bleeding complications, pneumonia). 0 to 48h: Dose needed of anti-shivering medication, level of sedation (RASS, GCS and BIS), safety laboratory including specific coagulation parameters and monitoring of cerebral auto-regulation including cNIRS and BIS.

CONTACTS AND LOCATIONS:
Overall Officials: Sven Poli, Dr. med., Principal Investigator — University Hospital Heidelberg
Locations (1):
- Stroke Unit, Dept. of Neurology, University Hospital Heidelberg, Heidelberg, Germany